CLINICAL TRIAL: NCT01247740
Title: A Prospective, Controlled, Randomized, Blinded, Parallel Group Multicentre Study on the Safety and Efficacy of a Convenience Three-chamber Bag for Parenteral Nutrition in Post-operative Patients After Abdominal Surgery Versus a Compounded Monobag
Brief Title: Comparison of Three-chamber-bag Versus Compounded Bag
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC-G-H-0805
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Parenteral Nutrition for Patients With Proven Insufficient Enteral Resorption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): three chamber bag for parenteral nutrition containing lipids, glucose, amino acids and electrolytes
  Interventions: Drug: NuTRIflex Lipid peri
- 2 (Active Comparator): compounded monobag including lipids, glucose, amino acids and electrolytes
  Interventions: Drug: compounded monobag

INTERVENTIONS:
Drug: NuTRIflex Lipid peri — parenteral nutrition
  Arms: 1
Drug: compounded monobag — parenteral nutrition
  Arms: 2

SUMMARY:
The purpose of the study is to investigate the efficacy and safety of a convenient 3-chamber-bag containing aminoacids, glucose and lipid emulsion (LCT/MCT 20%) compared to a conventionally compounded monobag for parenteral nutrition.

ELIGIBILITY:
Inclusion: •Patients considered for elective open abdominal surgery

* Male and female patients ≥18 and <85 years of age
* Indication for total parenteral nutrition therapy: for 6 consecutive days
* NRS ≥3
* Ability and willingness to give voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the Institutional Review Board (IRB) prior to all evaluations, and to comply with the requirements of the study

Exclusion: Major criteria:

* Body weight < 50 kg or > 70 kg
* Laparoscopic surgery
* Seriously ill patients in need of high energy nutrition support (i. e. > 2100 Kcal/day)
* Hepatic surgery
* Surgery with estimated blood loss >1000ml
* Participation in a clinical study with an investigational drug or an investigational medical device within one month prior to the start of study
* Receiving regular parenteral nutrition within 7 days before the onset of study
* General contraindications for parenteral nutrition (acidosis of various geneses, untreated disorders of electrolyte and fluid balance, hyperhydration, acute pulmonary edema, inadequate cellular oxygen supply)
* General contraindications for infusion therapy such as acute pulmonary oedema, hyperhydration and decompensated cardiac insufficiency, acute stroke
* Known hypersensitivity to egg-, soy-, and peanut proteins or any of the ingredients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Course of prealbumin (from day 1 to day 7) | 7 days

SECONDARY OUTCOMES:
clinical outcome parameters, haematology, liver function, blood biochemistry and electrolytes, coagulation function | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jianchun Yu, Prof., Principal Investigator — Peking Union Medical College Hospital,Department of Gastrointestinal Surgery
Locations (1):
- Peking Union Medical College Hospital,Department of Gastrointestinal Surgery, Beijing, China